CLINICAL TRIAL: NCT02587676
Title: Changes in the Hardness of Resilient Denture Liners Embedded in Maxillary Complete Dentures and Their Association With Patient Characteristics
Brief Title: Deterioration of Resilient Denture Liners and Patient Characteristics
Status: Completed | Type: Observational
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Yasuhiko Kawai, Professor Dr.Yasuhiko kawai, Nihon University
Other Study IDs: EC13-006
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Xerostomia; Menopause; Kidney Disease
MeSH Terms: conditions — Xerostomia; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- denture liners: Evatouch Super (EVA; Neo Dental Chemical products, Washington, USA), GC RELINE (GCR; GC Dental Products Corp, Tokyo, Japan), Mucopren soft (MCP; Kettenbach GmbH & Co KG, California, USA) Soften (SFT; KAMEMIZU CHEM, Osaka, Japan), FD Soft (FDS; KAMEMIZU CHEM, Osaka, Japan), and Bio Liner (BIO; Nissin Dental Products, Kyoto, Japan).
  Interventions: Other: Evatouch Super

INTERVENTIONS:
Other: Evatouch Super — The deterioration of RDLs may differ between in vitro conditions and the conditions encountered in denture wearers. We conducted an in vivo study to investigate how resilient denture liners (RDLs) changed in hardness when embedded in complete maxillary dentures worn by patients for one month in a clinical setting. We hypothesized that the hardness one month after application of the RDLs would be affected by the age, the condition of the saliva, the occlusal force, type of denture used, the patients habits related to smoking, drinking, wearing dentures while sleeping, and using a denture cleanser.
  Other Names: GC RELINE; Mucopren soft; Soften; FD Soft; Bio Liner

SUMMARY:
Thirty complete maxillary denture wearers were recruited after obtaining informed consent. One investigator measured the Shore D hardness of the commercially available RDLs using a Vesmeter®. The salivary flow rates and pH values and the occlusal force were measured for all patients before initiation of the study.

T-tests and Pearson's correlation coefficients were used for statistical analyses.

A p-value of <0.05 was considered statistically significant.

DETAILED DESCRIPTION:
1. Participants This study was approved by the Human Ethics Committee of Nihon University School of Dentistry, Matsudo (EC 13-006). Thirty wearers of complete maxillary dentures (12 men; mean age, 71.8 ± 9.2 years and 18 women; mean age, 70.2 ± 10.7 years) who visited the Department of Removable Prosthodontics at our institute were recruited for this study. The volunteers were enrolled only after they provided written informed consent. Complete maxillary denture wearers who had been treated with a tissue conditioner, RDLs, and denture adhesives were excluded. Before starting the clinical trial, the participants were asked about the following environmental factors in a questionnaire: smoking, drinking, denture wearing during sleeping, and denture cleanser usage.

   After specimen making, all participants were instructed to wear their dentures as per their normal routine.
2. Specimen Preparation A cylinder shapes six places with a 4-mm diameter and 2-mm depth , that was drilled into the inner surface of the denture base. Then, the RDL materials were mixed by each product, packed into the cavity, and polymerized at room temperature . The six commercial RDLs used in this study:Evatouch Super (EVA; Neo Dental Chemical products, Washington, USA), GC RELINE (GCR; GC Dental Products Corp, Tokyo, Japan), Mucopren soft (MCP; Kettenbach GmbH & Co KG, California, USA) Soften (SFT; KAMEMIZU CHEM, Osaka, Japan), FD Soft (FDS; KAMEMIZU CHEM, Osaka, Japan), and Bio Liner (BIO; Nissin Dental Products, Kyoto, Japan).

   Hardness was measured using a Vesmeter® (WaveCyber Corp, Saitama, Japan). When the probe, which included a built-in position sensor connected to a personal computer, was placed in a perpendicular orientation to an RDL, the indenter of the probe was depressed onto the RDL at a constant speed through electromagnetic power. Simultaneously, the path of the indenter was constantly traced by the position sensor. The computer processed electrical signals from the measuring device and calculated the Shore D hardness, which was the primary outcome in the present study. The same investigator measured the hardness at each appointment. The original hardness and the hardness at 1 month after oral exposure were used for analysis. Each specimen was measured five times, and the highest and lowest values were eliminated from the calculation of the mean representative value for each specimen. The specimens embedded in the dentures were measured on a hot plate to maintain the temperature at 37°C or as close to the oral temperature as possible.
3. Statistical Analyses Before other statistical analyses, the normality of the data was tested using the Kolmogorov - Smirnov test, and then parametric statistical methods were applied.Two-way repeated measures analysis of variance ( ANOVA ) with the material type (EVA, MCP, GCR, FDS, SFT, and BIO) and time period (baseline and one month after) as factors was used to assess changes in the hardness of the six RDLs over time. The Tukey-Kramer test was used as a post hoc test after the two-way repeated measures ANOVA .The effects of categorical variables such as sex, smoking, drinking, denture wearing during sleeping, and denture cleanser usage on the hardness of the RDLs were analyzed using a two-way ANOVA without a post hoc test; we were not interested in comparing each RDL but rather in analyzing the effects of categorical variables on the RDLs. The effects of continuous variables, including age, salivary flow rate, and occlusal force, were analyzed using Pearson's correlation coefficients. All statistical analyses were performed using IBM® SPSS® Statistics 21 (IBM, Armonk, NY, USA). A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* wearing maxillary complete dentures

Exclusion Criteria:

* had been treated with a tissue conditioner, RDLs, and denture adhesives were excluded
* showed obvious cognitive impairment
* could not understand written or spoken Japanese

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient of wearing complete maxillary dentures who visited the Department of Removable Prosthodontics at our institute were recruited for this study.
  The volunteers were enrolled only after they provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
hardness | 10 min
  Denture liners's hardness was measured using a Vesmeter® (WaveCyber Corp, Saitama ,Japan) at the out of oral cavity.

SECONDARY OUTCOMES:
Salivary flow test(Unstimulated saliva) | 5 min
  The participants were instructed to sit in an upright position with their heads inclined forward, which facilitated saliva collection at the floor of the mouth and overflow from the lip. The saliva was allowed to drip into a measuring cup for 5 min, and the flow rate was calculated in mL/min .
Salivary flow test(Stimulated saliva) | 2min
  The participants were instructed to chew a piece of paraffin gum until it became soft. The first collection of saliva was swallowed, the timer was set, and chewing was continued for another 2 min .The participants spat out the saliva at short intervals into a measuring cup. The participants were instructed not to eat anything (drinking water was allowed), smoke, or take snuff at least two hours before the tests.

OTHER OUTCOMES:
pH measurement | 5 min
  The pH values of the resting and stimulated saliva were obtained using a pH testing device (pH Spear, Eutech Instruments Pte Ltd, Ayer Rajah Crescent, Singapore). The investigator dipped the electrode approximately 2 to 3 cm into the saliva in a measuring cup and recorded the digitally obtained value.
Occlusal force measurement | 5 min
  A GM10 occlusal force meter (Nagano Keiki, Tokyo, Japan) was used to measure the occlusal force. The maximum occlusal force applied by the functioning left and right first molars was measured three times, and the mean was used as a representative value.
Questionnaire | 10 min
  Before starting the clinical trial, the participants were asked about the following environmental factors in a questionnaire: smoking, drinking, denture wearing during sleeping, and denture cleanser usage.

CONTACTS AND LOCATIONS:
Overall Officials: Akina Ogawa, Principal Investigator — Depertment of removable prosthodontics Nihon University School of Dentistry at Matsudo

REFERENCES:
- [Background] Kimoto S, So K, Yamamoto S, Ohno Y, Shinomiya M, Ogura K, Kobayashi K. Randomized controlled clinical trial for verifying the effect of silicone-based resilient denture liner on the masticatory function of complete denture wearers. Int J Prosthodont. 2006 Nov-Dec;19(6):593-600. PMID 17165299